CLINICAL TRIAL: NCT00789061
Title: Applying Proton Pump Inhibitor to Prevent and Treat Acute Fluctuating Hearing Loss in Patients With SLC26A4 Mutation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: WU CHEN-CHI
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 950805
Record Dates: First submitted 2007-07-08; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Hearing Loss
Keywords: Acute hearing loss in patients with SLC26A4 mutations
MeSH Terms: conditions — Hearing Loss | interventions — Proton Pump Inhibitors; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Proton pump inhibitor — One dosage/day/year
  Other Names: Taquidine,Lansoprazole

SUMMARY:
Disequilibrium between acid and base in the inner ear was suggested to be an important factor leading to hearing impairment associated with SLC26A4 mutations. For acid-base homeostasis in the inner ear, gastric-type proton pumps might demonstrate antagonistic effects to pendrin, the protein encoded by SLC26A4. To investigate whether proton pump inhibitors might prevent or treat acute fluctuating hearing loss related to SLC26A4 mutations, we launch the current double-blind randomized clinical trial.

DETAILED DESCRIPTION:
Hereditary hearing loss is the most common inherited sensory defect, affecting about 1 per 1000 children. With the advances in molecular genetics, the nature of hereditary hearing loss has started to be unraveled. A plethora of deafness genes were discovered in the past years, and among them certain genetic mutations were noted to be extraordinarily popular in the hearing-impaired population. For example, mutations in the SLC26A4 gene have been documented with high prevalence in a variety of ethnic backgrounds, including Caucasians, Japanese and Han Chinese.

The two specific clinical features of patients with SLC26A4 mutations are inner ear malformations and fluctuating hearing loss. For decades, the latter has constituted a treatment difficulty for pediatric otologists, because traditional regimens, such as steroid or intracranial-pressure-lowering-medication, usually could not achieve satisfactory and predictable outcomes. Nevertheless, as basic researches in recent years began to shed light on the pathogenesis of hearing loss from SLC26A4 mutations, novel strategies could be developed based on some of these crucial findings. For instance, disequilibrium between acid and base in the inner ear was reported to be an important factor leading to deafness in SLC26A4 knock-out mice. And for acid-base homeostasis in the inner ear, proton pumps were found to demonstrate antagonistic effects to pendrin, the protein encoded by SLC26A4. Consequently, regimens which can modulate the function of proton pumps, like proton pump inhibitors, might be a good choice to prevent or treat acute or chronic hearing loss related to SLC26A4 mutations or degenerative dysfunction.

Corresponding to this postulation, clinically we experienced significant recovery of hearing loss in several patients with SLC26A4 mutations who suffered from acute fluctuating hearing loss which was refractory to traditional treatment. In some cases, acute hearing loss recurred after the medication was discontinued. Therefore, we launch the current clinical trial to investigate the efficacy of proton pump inhibitor in preventing and treating acute hearing loss in patients with SLC26A4 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with homozygous or heterozygous SLC26A4 mutations
* Patients with acute hearing loss

Exclusion Criteria:

* Patients who do not fulfill both of the above criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-03 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Decrease in attack frequency or improvement of hearing loss | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chuan-Jen Hsu, MD, Study Director — Department of Otolaryngology, National Taiwan University Hospital; Chen-Chi Wu, MD, Principal Investigator — Department of Otolaryngology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan